CLINICAL TRIAL: NCT03963804
Title: Objective Brain Function Assessment of mTBI From Initial Injury to Rehabilitation in Concussion
Brief Title: Objective Brain Function Assessment of mTBI/Concussion
Acronym: CAS13-25
Status: Completed | Type: Observational
Sponsor: BrainScope Company, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 31-Ahead
Record Dates: First submitted 2019-05-21; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Brain Injuries, Traumatic; Concussion, Mild; Concussion, Intermediate; Concussion, Severe; Concussion, Brain
Keywords: Concussion; Mild Traumatic Brain Injury; Sport Related Concussion; Non-Sport Related Concussion
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Injured and Matched Control Subject Pool: Injured subjects consist of subjects who are head injured and meet the inclusion/exclusion criteria. Injured subjects will be tested within 72 hours (3 days) of injury and at specified time points post injury. Matched control subjects will be tested at the same time intervals as the injured subject. BrainScope Battery will be performed at each time point and consists of the following components: brain electrical activity (EEG), neurocognitive performance assessment, ocular motor assessment, and clinical symptoms/assessments.
  Interventions: Device: BrainScope Ahead 300iP
- Healthy Volunteer Subject Pool: This subject pool will consist of uninjured (not head injured) subjects and will be tested at a single time point. These subjects will perform the same BrainScope Battery as the injured and matched control subjects.
  Interventions: Device: BrainScope Ahead 300iP

INTERVENTIONS:
Device: BrainScope Ahead 300iP — The BrainScope Battery evaluation will consist of 4 tests to aid in the assessment of concussion: History, Physical, signs and symptoms (SAC, SCAT5), Electrophysiological Function; Neurocognitive Performance Assessment and Ocular Motor Assessment. BrainScope Ahead 300iP will be used to perform EEG and Cognitive assessments.

SUMMARY:
This study (Part 3) is designed to build a database including EEG, neurocognitive performance, clinical symptoms, history and other relevant data, which will be used to derive a multimodal EEG based algorithm for the identification of concussion and tracking of recovery.

DETAILED DESCRIPTION:
Injured/concussed subjects will be studied at time of injury, and at 3 follow-up time points following injury. Subjects will come from the sports and other populations of concussed individuals. They will be matched with controls i.e. not head injured subjects who will also undergo the same set of tests and the same time intervals as the injured subjects. An additional pool of uninjured (not head injured) subjects will be collected who will be assessed at a single time point. This data will be used to populate a database for the purpose of deriving a multimodal concussion index.

ELIGIBILITY:
Inclusion Criteria:

For Injured subjects:

1. Having sustained a traumatic closed head injury within 72 hours (3 days) from time of injury at time of BrainScope assessment;
2. GCS 13-15 at time of BrainScope assessment;
3. No hospital admission due to either head injury or collateral injuries for >24 hours.

For Matched Controls:

1. GCS 15 at time of BrainScope assessment;
2. No prior history of concussion or TBI in the last year.

Exclusion Criteria:

1. Previously enrolled in the BrainScope CAS Studies;
2. Current CNS active prescription medications taken daily, with the exception of medications being taken for the treatment of Attention Deficit Disorder (ADD) or Attention Deficit Hyperactivity Disorder (ADHD);
3. Forehead, scalp or skull abnormalities that prevents headset application or EEG data collection;
4. History of brain surgery or neurological disease;
5. Pregnant women;
6. Subjects who do not speak English (non-English speaking parents are allowed to consent so long as translation of the consent form in their native language is available);
7. Acute intoxication;
8. Evidence of illicit drug usage;

For Injured subjects:

1. Loss of consciousness ≥ 20 minutes related to the concussion injury;
2. Active fever defined as greater than 100ºF or 37.78ºC at time of BrainScope assessment;
3. Evidence of abnormality visible on Computerized Tomography (CT) of the head related to the traumatic event (Note: neuroimaging is not required for enrollment).

For Matched Controls:

1. Any focal neurological signs including aphasia, apraxia, diplopia, facial droop, dysarthria/slurred speech;
2. History of Motor Vehicle Accident (MVA) requiring an Emergency Department visit within the past 1 year.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Approximately 490 Injured, Matched Control and Healthy Volunteer subjects will be recruited from high schools, college universities, concussion clinics and emergency rooms.
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Derivation of algorithm for Likelihood of being concussed using multimodal inputs | 6 months for data acquisition, with each patient studied from time of injury to 45 days after RTP
  Create a database of all assessments including brain electrical activity (EEG features including all frequency bands and measures (power, connectivity,complexity), neurocognitive performance tests scores (throughput measures), balance, and clinical/symptom assessments (SCAT5), to support derivation of a multimodal brain function/concussion index. (NOTE: All EEG and Neurocognitive features are expressed as z-scores relative to age expected normal values to enable combination)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Prichep, Ph.D., Study Director — BrainScope Company, Inc.
Locations (4):
- United States (4):
  - University of Arkansas, Fayetteville, Arkansas
  - University of Miami, Miami, Florida
  - Michigan State University, East Lansing, Michigan
  - University of Rochester, Rochester, New York

REFERENCES:
- [Derived] Covassin T, McGowan AL, Bretzin AC, Anderson M, Petit KM, Savage JL, Katie SL, Elbin RJ, Pontifex MB. Preliminary investigation of a multimodal enhanced brain function index among high school and collegiate concussed male and female athletes. Phys Sportsmed. 2020 Nov;48(4):442-449. doi: 10.1080/00913847.2020.1745717. Epub 2020 Mar 31. PMID 32228157